CLINICAL TRIAL: NCT06767839
Title: The Effect of Different Electrotherapy Interventions on Pain and Hand Function in Young Individuals With Neck Pain: a Randomized Controlled Double-blind Trial
Brief Title: The Effect of Electrotherapy on Young Individuals With Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Betül Söylemez, Lecturer, PT.MSc., Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO 2023/97
Record Dates: First submitted 2024-12-17; First posted 2025-01-10 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Neck Pain
Keywords: neck pain; electrotherapy; TENS; HVPGS
MeSH Terms: conditions — Neck Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The sample of the study is Burdur Health Services Vocational School students with neck pain. Participants will be assigned to 3 intervention groups by stratified randomization. The strata are age and gender.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group of Transcutaneous Electrical Nerve Stimulation (TENS) (Experimental): Participants assigned to this group will receive TENS for 20 minutes each session for a total of 20 sessions.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation
- Group of High Voltage Pulsed Galvanic Stimulation (HVPGS) (Experimental): Participants assigned to this group will receive HVPGS for 20 minutes each session for a total of 20 sessions.
  Interventions: Other: High Voltage Pulsed Galvanic Stimulation
- Group of sham (Sham Comparator): Individuals assigned to this group will be started on TENS current for a total of 20 sessions, each session lasting 20 minutes, but the current will be reduced and turned off after 1 minute. It will be explained to the individuals that this current is applied at a subthreshold level.
  Interventions: Other: Sham TENS

INTERVENTIONS:
Other: Transcutaneous Electrical Nerve Stimulation — The current parameters for the TENS to be applied in the study were determined as 100 Hz, 100 microsecond pulse duration, and asymmetric biphasic waveform. The current intensity will be increased until the person feels a tingling sensation and will be applied for a total of 20 minutes. Two superficial electrodes will be placed to cover the application area to create an effect in deep tissue.
  Other Names: TENS
  Arms: Group of Transcutaneous Electrical Nerve Stimulation (TENS)
Other: High Voltage Pulsed Galvanic Stimulation — YVKGS is a monophasic waveform current with double peaks, short pulse duration and a voltage higher than 100 Volts, the frequency of which can be adjusted optionally. In the study, the current parameters of YVKGS were determined as a frequency of 100 Hz, continuous pulse, double peak monophasic waveform. The current intensity will be applied for 20 minutes at the voltage at which the person feels a tingling sensation. Two superficial electrodes will be placed to cover the application area to create an effect in deep tissue.
  Other Names: HVPGS
  Arms: Group of High Voltage Pulsed Galvanic Stimulation (HVPGS)
Other: Sham TENS — The current will be applied to the sham TENS group with the same parameters as the TENS group, and will be reduced and turned off after a while. In TENS application, people normally report that they no longer feel tingling after a few minutes of starting the application. Therefore, it will be explained to the sham TENS group that this situation is normal, and that they no longer feel tingling because they have become accustomed to the applied current.
  Arms: Group of sham

SUMMARY:
The aim of this clinical study was to investigate the effects of different electrotherapy interventions on pain and hand function in young individuals with neck pain.

The main question that the study aimed to answer is: are two different electrotherapy interventions superior to each other for pain and hand function? Participants will be assigned to either transcutaneous electrical nerve stimulation, high-voltage pulsed galvanic stimulation, or placebo. Participants will receive a total of 20 sessions of electrotherapy intervention, 20 minutes per day, 3 days a week. Participants will be evaluated before the intervention, after 1 session, and 1 week after the completion of the 20-session intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-30 years old
* Complaining of neck pain
* Volunteering to participate in the study

Exclusion Criteria:

* Having received any anti-inflammatory treatment in the last 3 months
* Having received any physical therapy and rehabilitation treatment in the last 3 months
* Doing regular exercise
* Not attending work sessions

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | From enrollment to the end of treatment at 7 weeks
  The Visual Analog Scale is a 10-centimeter (cm) scale, with 0 being defined as "no pain" and 10 as "unbearable pain." It is a valid and reliable method for assessing the severity of musculoskeletal pain and is frequently used in clinical studies. In a study conducted on patients with chronic musculoskeletal pain, a VAS value of less than 3.4 cm was classified as mild pain, a VAS value between 3.5 and 7.4 cm was classified as moderate pain, and a VAS value greater than 7.5 cm was classified as severe pain.
Treshold Faradic Test | From enrollment to the end of treatment at 7 weeks
  Pain threshold measurement is performed by applying a surge faradic current with a frequency of 50 Hz and a transition time of 0.1-1 msec. The point at which the current is first felt is defined as the pain threshold. In this test, the active electrode is placed at the motor point of the relevant muscle, while the passive electrode can be placed in a more distal or proximal region.
Patient-Specific Functional Scale | From enrollment to the end of treatment at 7 weeks
  Patients are asked to list the three activities that cause the most difficulty with their neck pain. Each activity is then scored from 0 (unable to perform the activity) to 10 (able to perform the activity at the same level as before the onset of symptoms).
Core Outcome Meassure Index-Neck | From enrollment to the end of treatment at 7 weeks
  It is a symptom-specific measurement tool that includes all the parameters that need to be evaluated in patients with low back pain (pain, function, quality of life, disability), and has the advantages of being short and easy to apply. It consists of six questions and each question is scored between 0 and 10. Higher scores indicate worse results.

SECONDARY OUTCOMES:
Nine-Hole Peg Test | From enrollment to the end of treatment at 7 weeks
  It is a standardized, valid and reliable test that measures upper extremity functions and motor speed, consisting of nine cylindrical wooden sticks and a board with nine round holes. Individuals are asked to quickly take 9 wooden sticks from the box they are in, place them in the holes randomly without observing the order, quickly take them out of the holes without waiting and place them back in the box. The total time that elapses while the individuals insert and remove the sticks from the holes is recorded with a stopwatch in seconds.
Gross Grip Strength | From enrollment to the end of treatment at 7 weeks
  Gross grip strength will be measured with a Jamar® digital hand dynamometer. The gross grip strength measurement will be performed in the standard measurement position recommended by the American Hand Therapists Association, with the patient sitting in a chair without elbow support, the arm in adduction and neutral rotation, the elbow in 90-degree flexion, and the forearm and wrist in a neutral position. The test will be repeated 3 times. The average of the 3 tests will be taken.
Pinch Grip Strength | From enrollment to the end of treatment at 7 weeks
  Pinch grip strength will be measured with a Jamar® digital pinchmeter. The pinch grip strength measurement position will be performed with the patient sitting in a chair without elbow support, the arm in adduction and neutral rotation, the elbow in 90 degrees flexion, the forearm in 90 degrees supination, and the wrist in a neutral position. The test will be repeated 3 times. The average of the 3 tests will be taken.
Upper Extremity Strenght | From enrollment to the end of treatment at 7 weeks
  The strength of individuals' shoulder flexor, extensor, abductor, adductor and rotator muscles, elbow flexor and extensor muscles, wrist flexor and extensor muscles will be evaluated with a sphygmomanometer. The evaluation will be carried out with the protocol of the person being measured applying maximum force against the device while the person measuring holds the sphygmomanometer steady.
Semmes-Weinstein Monofilament Test | From enrollment to the end of treatment at 7 weeks
  It is a test used to evaluate light touch sensation in individuals. Monofilaments contain different values from 1.65 to 6.65. Monofilaments between 1.65 and 2.83 are interpreted as normal sensation, while an increase in the perceived thickness indicates a sensory defect. The test will be applied to the C3-C8 dermatomes on both upper extremities. The evaluation will start with the 2.83 monofilament, which is considered optimal, and 3 strokes, each lasting 3 seconds, will be applied to each point with the monofilament. Individuals will be asked to give the answer "I felt it". If individuals respond, a lower monofilament will be applied, and if no response is received, a higher monofilament will be applied and the test will be continued.
Cervical Endurance Test | From enrollment to the end of treatment at 7 weeks
  To assess the endurance of the cervical flexors, individuals perform cervical flexion while lying on their back in a chin position, and the time they maintain this position is recorded in seconds. To assess the endurance of the cervical extensors, individuals attempt to maintain a neutral neck position while lying on their stomach with their head hanging off the bed, and the time they maintain this position is recorded in seconds. The test is terminated when the head position changes in the direction of flexion or extension, or when individuals want to stop the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parazza S, Vanti C, O'Reilly C, Villafane JH, Tricas Moreno JM, Estebanez De Miguel E. The relationship between cervical flexor endurance, cervical extensor endurance, VAS, and disability in subjects with neck pain. Chiropr Man Therap. 2014 Mar 3;22(1):10. doi: 10.1186/2045-709X-22-10. PMID 24581272
- [Background] Olson LE, Millar AL, Dunker J, Hicks J, Glanz D. Reliability of a clinical test for deep cervical flexor endurance. J Manipulative Physiol Ther. 2006 Feb;29(2):134-8. doi: 10.1016/j.jmpt.2005.12.009. PMID 16461172
- [Background] Bell-Krotoski JA, Fess EE, Figarola JH, Hiltz D. Threshold detection and Semmes-Weinstein monofilaments. J Hand Ther. 1995 Apr-Jun;8(2):155-62. doi: 10.1016/s0894-1130(12)80314-0. PMID 7550627
- [Background] Raji P, Ansari NN, Naghdi S, Forogh B, Hasson S. Relationship between Semmes-Weinstein Monofilaments perception Test and sensory nerve conduction studies in Carpal Tunnel Syndrome. NeuroRehabilitation. 2014;35(3):543-52. doi: 10.3233/NRE-141150. PMID 25238864
- [Background] Mannion AF, Porchet F, Kleinstuck FS, Lattig F, Jeszenszky D, Bartanusz V, Dvorak J, Grob D. The quality of spine surgery from the patient's perspective. Part 1: the Core Outcome Measures Index in clinical practice. Eur Spine J. 2009 Aug;18 Suppl 3(Suppl 3):367-73. doi: 10.1007/s00586-009-0942-8. Epub 2009 Mar 25. PMID 19319578
- [Background] Stevens A, Koke A, van der Weijden T, Beurskens A. The development of a patient-specific method for physiotherapy goal setting: a user-centered design. Disabil Rehabil. 2018 Aug;40(17):2048-2055. doi: 10.1080/09638288.2017.1325943. Epub 2017 May 13. PMID 28504014
- [Background] Boonstra AM, Schiphorst Preuper HR, Balk GA, Stewart RE. Cut-off points for mild, moderate, and severe pain on the visual analogue scale for pain in patients with chronic musculoskeletal pain. Pain. 2014 Dec;155(12):2545-2550. doi: 10.1016/j.pain.2014.09.014. Epub 2014 Sep 17. PMID 25239073
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Background] Yalcinkaya G, Kara B, Arda MN. Cross-cultural adaptation, reliability and validity of the Turkish version of Patient-Specific Functional Scale in patients with chronic neck pain. Turk J Med Sci. 2020 Jun 23;50(4):824-831. doi: 10.3906/sag-1905-91. PMID 32233180
- [Background] Dissanayaka TD, Pallegama RW, Suraweera HJ, Johnson MI, Kariyawasam AP. Comparison of the Effectiveness of Transcutaneous Electrical Nerve Stimulation and Interferential Therapy on the Upper Trapezius in Myofascial Pain Syndrome: A Randomized Controlled Study. Am J Phys Med Rehabil. 2016 Sep;95(9):663-72. doi: 10.1097/PHM.0000000000000461. PMID 26945216
- [Background] Chen PY, Cheen JR, Jheng YC, Wu HK, Huang SE, Kao CL. Clinical applications and consideration of interventions of electrotherapy for orthopedic and neurological rehabilitation. J Chin Med Assoc. 2022 Jan 1;85(1):24-29. doi: 10.1097/JCMA.0000000000000634. PMID 34643619
- [Background] Acedo AA, Luduvice Antunes AC, Barros dos Santos A, Barbosa de Olveira C, Tavares dos Santos C, Colonezi GL, Fontana FA, Fukuda TY. Upper trapezius relaxation induced by TENS and interferential current in computer users with chronic nonspecific neck discomfort: An electromyographic analysis. J Back Musculoskelet Rehabil. 2015;28(1):19-24. doi: 10.3233/BMR-140482. PMID 24867904
- [Background] Alsalameh AM, Harisi MJ, Alduayji MA, Almutham AA, Mahmood FM. Evaluating the relationship between smartphone addiction/overuse and musculoskeletal pain among medical students at Qassim University. J Family Med Prim Care. 2019 Sep 30;8(9):2953-2959. doi: 10.4103/jfmpc.jfmpc_665_19. eCollection 2019 Sep. PMID 31681674
- [Background] Xie Y, Szeto G, Dai J. Prevalence and risk factors associated with musculoskeletal complaints among users of mobile handheld devices: A systematic review. Appl Ergon. 2017 Mar;59(Pt A):132-142. doi: 10.1016/j.apergo.2016.08.020. Epub 2016 Sep 11. PMID 27890121
- [Background] Özünlü Pekyavaş, N. , Bastug Yuruk, O. & Saygılı, F. (2020). Artan Mobil Teknoloji Kullanımının Yol Açtığı Ağrı Sendromu: "Text Neck" . Adnan Menderes Üniversitesi Sağlık Bilimleri Fakültesi Dergisi , 4 (3) , 251-257 .
- [Background] Johnston V, Jull G, Darnell R, Jimmieson NL, Souvlis T. Alterations in cervical muscle activity in functional and stressful tasks in female office workers with neck pain. Eur J Appl Physiol. 2008 Jun;103(3):253-64. doi: 10.1007/s00421-008-0696-8. Epub 2008 Feb 22. PMID 18293008
- [Background] Blozik E, Laptinskaya D, Herrmann-Lingen C, Schaefer H, Kochen MM, Himmel W, Scherer M. Depression and anxiety as major determinants of neck pain: a cross-sectional study in general practice. BMC Musculoskelet Disord. 2009 Jan 26;10:13. doi: 10.1186/1471-2474-10-13. PMID 19171034